CLINICAL TRIAL: NCT06120569
Title: Evaluate the Role of Soleus Muscle Exercise in Glycaemic Control in Diabetic Kidney Disease Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nora Hussein Kamal (Other)
Responsible Party: Sponsor-Investigator, Nora Hussein Kamal, Internal medicine doctor, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Soleus ms exercise in diabetis
Record Dates: First submitted 2023-10-19; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Diabetic Kidney Disease
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Soleus muscle exercise in diabetes (Experimental): Soleus muscle decrease blood glucose
  Interventions: Device: Soleus ms exercise
- Decrease glucose level by soleus exercise (Experimental): Soleus ms exercise in decrease blood glucose
  Interventions: Device: Soleus ms exercise

INTERVENTIONS:
Device: Soleus ms exercise — Soleus muscle exercise before and after eating by half an hour

SUMMARY:
Evaluate the role of Soleus muscle exercise in management diabetic kidney disease

DETAILED DESCRIPTION:
management of diabetic kidney disease. To enhance their glycemic control, diabetic patients are advised to perform 150 minutes per week of moderate-to-vigorous aerobic activity Diabetic patients with regular physical activity have reduced daily insulin dose with more glycemic control. In addition to glycemic control, it has also been postulated that the addition of brief intervals of high intensity, sprint -type exercise to aerobic exercise can decrease the risk of late nocturnal hypoglycemic episodes Marc T. Hamilton et al., 2022, reported that the human soleus muscle could raise local oxidative metabolism to high levels for hours without fatigue, during a type of soleus-dominant activity while sitting (soleus push up exercise), even in unfit volunteers. They reported that soleus push up exercise can improve systemic VLDL-triglyceride and glucose homeostasis by a large magnitude, e.g., 52% less postprandial glucose excursion (∼50 mg/dL less between ∼1 and 2 h) with 60% less hyperinsulinemia. Muscle biopsies revealed there was minimal glycogen use. This can be explained that the soleus doesn't rely completely on intramuscular glycogen, Instead, it uses a mixture of fuels from glucose and lipoproteins.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18-60 yrs.,
* patients with Diabetic kidney disease, not on dialysis
* with stabilized diabetic treatment regimen for 3 months before participating in the study

Exclusion Criteria:

* advanced osteoarthritis of lower limb joints
* advanced poly neuropathic patients
* CKD type V on dialysis
* Diabetic Foot
* hemophilia
* bleeding tendency
* AKI
* other causes of chronic kidney disease
* patients refuse to participate in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-09-18 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
HbA1C less than 7% | One year
  Improve HbA1c by soleus muscle exercise

SECONDARY OUTCOMES:
ratio of albumin (mcg/L) to creatinine (mg/L)ratio | One year
  Improve alb /creatinine ratio

CONTACTS AND LOCATIONS:
Overall Officials: Samir Kamal, Ass prof, Study Director — Superviosor

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Pudmed — http://pubmed.ncbi.nlm.nih.gov/30559231/